CLINICAL TRIAL: NCT01154023
Title: Behavioral Intervention for Insomnia in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl T. Hayden VA Medical Center (U.S. Federal Agency)
Responsible Party: Dana R. Epstein, Carl T. Hayden Veterans Affairs Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R29NR004951 (NIH)
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Sleep Initiation and Maintenance Disorders; Behavior Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- stimulus control therapy (Experimental): Focuses on strengthening the bed and bedroom as cues for sleepiness and sleep, weaken them as cues for arousal, and developing a consistent sleep-wake pattern
  Interventions: Behavioral: stimulus control therapy, sleep restriction therapy, multi-component treatment (stimulus control therapy, sleep restriction therapy)
- sleep restriction therapy (Experimental): Sleep restriction therapy consolidates sleep by restricting the amount of time spent in bed and limiting sleep to a specific time period .
  Interventions: Behavioral: stimulus control therapy, sleep restriction therapy, multi-component treatment (stimulus control therapy, sleep restriction therapy)
- multi-component intervention (Experimental): Combines stimulus control and sleep restriction: strengthen the bed and bedroom as cues for sleepiness and sleep, weaken them as cues for arousal, develop a consistent sleep-wake pattern, consolidate sleep by restricting the amount of time spent in bed and limit sleep to a specific time period
  Interventions: Behavioral: stimulus control therapy, sleep restriction therapy, multi-component treatment (stimulus control therapy, sleep restriction therapy)

INTERVENTIONS:
Behavioral: stimulus control therapy, sleep restriction therapy, multi-component treatment (stimulus control therapy, sleep restriction therapy) — Treatment was given weekly for 6 weeks. Sessions 1 - 4 were in a group format. Session 5 & 6 were delivered individually by phone.

SUMMARY:
The purpose of the study was to evaluate and compare the efficacy of single interventions (stimulus control instructions, sleep restriction therapy) and multi-component intervention (stimulus control instructions and sleep restriction therapy) for chronic insomnia in community dwelling older adults. The subjects were randomly assigned to one of four conditions: stimulus control instructions, sleep restriction therapy, multi-component treatment (stimulus control instructions and sleep restriction therapy), or measurement control.

ELIGIBILITY:
Inclusion Criteria:

* 55 years or older
* Sleep onset or maintenance insomnia of 45 minutes or more per night for at least 3 nights per week as ascertained through 14 days of sleep diaries
* Insomnia duration of at least 6 months
* Impaired daytime functioning as a consequence of insomnia

Exclusion Criteria:

* Psychopathology evidenced by the Brief Symptom Inventory Global Severity Index T score >60
* Cognitive impairment as ascertained by the Mini-Mental State Exam score < 27
* Current psychotherapy or medical treatment for major depression or other psychopathology
* Current and regular use of over-the-counter medication or prescription medication for sleep (verified through urinalysis), or any medication affecting sleep
* Major physical or mental illness directly related to the onset and course of insomnia
* Substance abuse problem ascertained per interview
* Suspicion of sleep apnea as determined by an Epworth Sleepiness Scale score of 11 or greater, a respiratory disturbance index of > 15 as established through in-home overnight use of the EdenTec Model 3711 Digital Recorder, and interview with a significant other, if available
* Restless leg syndrome, periodic limb movement disorder, or circadian rhythm sleep disorders as determined through the participant interview and an interview with a significant other, if available.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2000-09; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
subjective sleep | 1 year
  daily sleep diaries were used for 2 weeks at each of the four measurement points, pre-treatment, post-treatment, 3 months and 1 year - called daily to voice mail service to avoid retrospective estimates of sleep

SECONDARY OUTCOMES:
insomnia severity | 1 year
  Insomnia Severity Index was used at the four measurement points (pre-treatment, post-treatment, 3 months, and 1 year) and also included the significant other version of the instrument

CONTACTS AND LOCATIONS:
Overall Officials: Dana R Epstein, PhD, RN, Principal Investigator — Carl T. Hayden VA

REFERENCES:
- [Derived] Epstein DR, Sidani S, Bootzin RR, Belyea MJ. Dismantling multicomponent behavioral treatment for insomnia in older adults: a randomized controlled trial. Sleep. 2012 Jun 1;35(6):797-805. doi: 10.5665/sleep.1878. PMID 22654199